CLINICAL TRIAL: NCT05120141
Title: Twelve Week Safety and Clinical Efficacy of Experimental Mouth Rinses
Brief Title: A Twelve Week Study of Experimental Mouth Rinses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CCSORC002549; CCSORC002549 (Other: Johnson & Johnson Consumer Inc. (J&JCI))
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Gingivitis; Plaque
MeSH Terms: conditions — Gingivitis; Plaque, Amyloid | interventions — American Dental Association

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Prototype 1 Mouth Rinse (Experimental): Participants will brush their teeth using soft bristled Toothbrush and Colgate Cavity Protection Toothpaste twice daily and rinse with 20 milliliters (mL) of the Prototype 1 Mouth Rinse for 30 seconds, twice a day following brushing on Day 0 under supervision and up to 12 weeks unsupervised at home.
  Interventions: Other: Colgate Cavity Protection Toothpaste; Other: American Dental Association (ADA) Ref Toothbrush; Other: Prototype 1 Mouth Rinse
- Prototype 2 Mouth Rinse (Experimental): Participants will brush their teeth using soft bristled Toothbrush and Colgate Cavity Protection Toothpaste twice daily and rinse with 20 mL of the Prototype 2 Mouth Rinse for 30 seconds, twice a day following brushing on Day 0 under supervision and up to 12 weeks unsupervised at home.
  Interventions: Other: Colgate Cavity Protection Toothpaste; Other: American Dental Association (ADA) Ref Toothbrush; Other: Prototype 2 Mouth Rinse
- Prototype 3 Mouth Rinse (Experimental): Participants will brush their teeth using soft bristled Toothbrush and Colgate Cavity Protection Toothpaste twice daily and rinse with 20 mL of the Prototype 3 Mouth Rinse for 30 seconds, twice a day following brushing on Day 0 under supervision and up to 12 weeks unsupervised at home.
  Interventions: Other: Colgate Cavity Protection Toothpaste; Other: American Dental Association (ADA) Ref Toothbrush; Other: Prototype 3 Mouth Rinse
- Listerine Cool Mint Mouth Rinse (Positive Control) (Active Comparator): Participants will brush their teeth using soft bristled Toothbrush and Colgate Cavity Protection Toothpaste twice daily and rinse with 20 mL of the Listerine Cool Mint Mouth rinse for 30 seconds, twice a day following brushing on Day 0 under supervision and up to 12 weeks unsupervised at home.
  Interventions: Other: Colgate Cavity Protection Toothpaste; Other: American Dental Association (ADA) Ref Toothbrush; Other: Listerine Cool Mint Mouth Rinse
- Hydroalcohol Mouth Rinse (Negative Control) (Active Comparator): Participants will brush their teeth using soft bristled Toothbrush and Colgate Cavity Protection Toothpaste twice daily and rinse with 20 mL of the Hydroalcohol Mouth Rinse for 30 seconds, twice a day following brushing on Day 0 under supervision and up to 12 weeks unsupervised at home.
  Interventions: Other: Colgate Cavity Protection Toothpaste; Other: American Dental Association (ADA) Ref Toothbrush; Other: Hydroalcohol Mouth Rinse

INTERVENTIONS:
Other: Colgate Cavity Protection Toothpaste — Participants will use Colgate Cavity Protection Toothpaste for brushing teeth twice daily.
Other: American Dental Association (ADA) Ref Toothbrush — Participants will use soft bristled Toothbrush for brushing teeth twice daily.
Other: Prototype 1 Mouth Rinse — Participants will use 20 mL of Prototype 1 Mouth Rinse for 30 seconds after brushing twice daily.
  Arms: Prototype 1 Mouth Rinse
Other: Prototype 2 Mouth Rinse — Participants will use 20 mL of Prototype 2 Mouth Rinse for 30 seconds after brushing twice daily.
  Arms: Prototype 2 Mouth Rinse
Other: Prototype 3 Mouth Rinse — Participants will use 20 mL of Prototype 3 Mouth Rinse for 30 seconds after brushing twice daily.
  Arms: Prototype 3 Mouth Rinse
Other: Listerine Cool Mint Mouth Rinse — Participants will use 20 mL of Listerine Cool Mint Mouth Rinse for 30 seconds after brushing twice daily.
  Arms: Listerine Cool Mint Mouth Rinse (Positive Control)
Other: Hydroalcohol Mouth Rinse — Participants will use 20 mL of Hydroalcohol Mouth Rinse for 30 seconds after brushing twice daily.
  Arms: Hydroalcohol Mouth Rinse (Negative Control)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of experimental mouth rinse formulations compared to a hydroalcohol control mouth rinse and a positive control mouth rinse for the reduction of gingivitis and plaque when used as an adjunct to tooth brushing during a twelve-week product usage period.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and follow the requirements and restrictions of the study (including willingness to use the assigned study products per instructions, availability on scheduled visit dates and likeliness of completing the clinical study) based upon research site personnel's assessment
* Evidence of a personally signed and dated informed consent document indicating the participant (or legally acceptable representative) has been informed of all pertinent aspects of the trial
* Able to read and understand the local language (participant is capable of reading the documents)
* Adequate oral hygiene (that is brush teeth daily and exhibit no signs of oral neglect)
* Adults, 18 to 60 years of age, in good general and oral health without any known allergy to commercial dental products or cosmetics
* Negative pregnancy urine tests (females of child-bearing potential only)
* Females of childbearing potential must be using a medically acceptable method of birth control for at least one month prior to Visit 1 and agree to continue using this method during their participation in the study
* A minimum of 20 natural teeth with scorable facial and lingual surfaces. Teeth that are grossly carious, extensively restored, orthodontically banded, abutments, exhibiting severe generalized cervical and/or enamel abrasion, or third molars will not be included in the tooth count
* A mean gingival index greater than or equal to (>=) 1.95 per the Modified Gingival Index at Baseline
* A mean plaque index >= 1.95 per the 6 site Turesky modification of the Quigley-Hein Plaque Index at Baseline
* Greater than or equal to 10 percent (%) bleeding sites at Baseline
* Absence of significant oral soft tissue pathology, excluding plaque-induced gingivitis, based on a visual examination and at the discretion of the Investigator
* Absence of moderate/advanced periodontitis based on a clinical examination and discretion of the dental examiner
* Absence of fixed or removable orthodontic appliance or removable partial dentures

Exclusion Criteria:

* History of significant adverse effects, including sensitivities or suspected allergies, following use of oral hygiene products such as toothpastes, mouth rinses and red food dye
* Dental prophylaxis within four weeks prior to Baseline visit
* More than three sites that have periodontal pockets depths measuring 5 millimeter (mm) in depth
* History of medical conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures
* Use of antibiotics, anti-inflammatory or anticoagulant therapy, phenytoin sodium or diphenylhydantoin, calcium channel blockers, cyclosporin A, immunostimulants/ immunomodulators during the study or within the one month prior to the Baseline exam.

Intermittent use of certain anti-inflammatory medication (ibuprofen, Aspirin) is acceptable at the discretion of the investigator

* Use of chemotherapeutic anti-plaque/anti-gingivitis products such as triclosan, essential oils, cetylpyridinium chloride, sodium fluoride with cetylpyridinium chloride (CPC), stannous fluoride, zinc or chlorhexidine digluconate containing mouth rinses and toothpastes within the four weeks prior to the Baseline exam
* Known allergy or sensitivity or history of significant adverse effects to any of the investigational product and/or product ingredients (or other ingredients in the products)
* Self-reported pregnancy or lactation (this criterion is due to oral tissue changes related to pregnancy and nursing which can affect interpretation of study results)
* Self-reported smokeless tobacco user including snuff, chewing tobacco, vaping and electronic (e)-cigarette usage
* Males with a pregnant partner or a partner who is currently trying to become pregnant
* Suspected alcohol or substance abuse (example., amphetamines, benzodiazepines, cocaine, marijuana, opiates)
* Significant unstable or uncontrolled medical condition which may interfere with a participant's participation in the study, including cancer, chronic kidney disease, chronic obstructive pulmonary disease (COPD), immunocompromised state (weakened immune system) from solid organ transplant, serious heart conditions, (such as heart failure, coronary artery disease, or cardiomyopathies) Sickle cell disease, Type 2 diabetes mellitus
* Participation in any clinical trial within 30 days of Screening visit
* Diagnosed Temporo-mandibular joint dysfunction/disorder
* Participants who wear bruxing devices, dental aligners, retainers
* Participants who were previously screened and ineligible or were randomized to receive investigational product
* Participants who are related to those persons involved directly or indirectly with the conduct of this study (that is, principal investigator, sub-investigators, study coordinators, other site personnel, employees of Johnson & Johnson subsidiaries, contractors of Johnson & Johnson, and the families of each)
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the participant inappropriate for entry into this study
* Coronavirus Disease 2019 (COVID-19) restrictions: a) History of a confirmed COVID-19 infection in the last 30 days; b) Contact with a COVID-19-infected person within 14 days prior to enrollment; c) Any international travel within 14 days prior to enrollment including members in the same household; d) Participants with self-reported symptoms within the past 2 weeks: i) Unexplained cough, shortness of breath/difficulty breathing, fatigue, body aches (headaches, muscle pain, stomach aches), conjunctivitis, loss of smell, loss of taste, poor appetite, nausea, vomiting, diarrhea, palpitations, fever or chest pain/tightness; ii) Temperature >= 38.0 degree Celsius (°C)/100.4 degree Fahrenheit (°F), measured by thermometer which is adjusted for core temperature; iii) Use of fever reducers within the past 2 days of each onsite visit

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2021-07-23 (Actual)

PRIMARY OUTCOMES:
Whole-mouth Mean Modified Gingival Index (MGI) Score After 12 Weeks of Product use | 12 weeks
  Gingivitis will be assessed by the MGI on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth: 0 (Normal [absence of inflammation]), 1 (Mild inflammation [slight change in color, little change in texture] of any portion of the entire gingival unit); 2 (Mild inflammation of the entire gingival unit); 3 (Moderate inflammation [moderate glazing, redness, edema, and/or hypertrophy] of the gingival unit); 4 (Severe inflammation [marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration] of the gingival unit).
Whole-mouth Mean Plaque Index (TPI) Score After 12 Weeks of Product use | 12 weeks
  Plaque area will be scored by the Turesky modification of the Quigley-Hein Plaque Index, on 6 surfaces (distobuccal, midbuccal and mesiobuccal, distolingual, midlingual and mesiolingual) of all scorable teeth, following disclosing: 0 (No Plaque); 1 (Separate flecks or discontinuous band of plaque around the gingival (cervical) margin); 2 (Thin (up to 1 millimeter [mm]), continuous band of plaque at the gingival margin); 3 (Band of plaque wider than 1mm but less than1/3 of the surface); 4 (Plaque covering 1/3 or more, but less than 2/3 of the surface); 5 (Plaque covering 2/3 or more of the surface).

SECONDARY OUTCOMES:
Whole-mouth Mean TPI Score After 1 and 4 Weeks of Product use | Weeks 1 and 4
  Plaque area will be scored by the Turesky modification of the Quigley-Hein Plaque Index, on 6 surfaces (distobuccal, midbuccal and mesiobuccal, distolingual, midlingual and mesiolingual) of all scorable teeth, following disclosing: 0 (No Plaque); 1 (Separate flecks or discontinuous band of plaque around the gingival (cervical) margin); 2 (Thin [up to 1 mm], continuous band of plaque at the gingival margin); 3 (Band of plaque wider than 1mm but less than1/3 of the surface); 4 (Plaque covering 1/3 or more, but less than 2/3 of the surface); 5 (Plaque covering 2/3 or more of the surface).
Whole-mouth Mean MGI Score After 4 Weeks of Product Use | 4 weeks
  Gingivitis will be assessed by the MGI on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth: 0 (Normal [absence of inflammation]), 1 (Mild inflammation [slight change in color, little change in texture] of any portion of the entire gingival unit); 2 (Mild inflammation of the entire gingival unit); 3 (Moderate inflammation [moderate glazing, redness, edema, and/or hypertrophy] of the gingival unit); 4 (Severe inflammation [marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration] of the gingival unit).
Whole-Mouth Mean Expanded Gingival Bleeding Index (EBI) Score at 4 and 12 Weeks of Product use | Weeks 4 and 12
  Bleeding will be assessed according to the EBI, 168 Sites. A periodontal probe with a 0.5 mm diameter tip will be inserted into the gingival crevice and swept from distal to mesial around the tooth at an angle of approximately 60 degrees, while in contact with the sulcular epithelium. Each of 6 gingival areas (distobuccal, mid-buccal, mesiobuccal, distolingual, mid-lingual, and mesiolingual) around each tooth will be assessed. After approximately 30 seconds, bleeding at each gingival unit will be recorded according to the following scale: 0 (Absence of bleeding after 30 seconds); 1 (Bleeding after 30 seconds); 2 (Immediate bleeding).
Percentage of Bleeding Sites, Based on the EBI Score at 4 and 12 Weeks of Product use | Weeks 4 and 12
  Percentage of bleeding sites will be calculated by taking the total number of sites with bleeding score greater than 0 divided by the total number of sites assessed for each participant. Bleeding will be assessed according to the Expanded Gingival Bleeding Index, 168 Sites. A periodontal probe with a 0.5 mm diameter tip will be inserted into the gingival crevice and swept from distal to mesial around the tooth at an angle of approximately 60 degrees, while in contact with the sulcular epithelium. Each of 6 gingival areas (distobuccal, mid-buccal, mesiobuccal, distolingual, mid-lingual, and mesiolingual) around each tooth will be assessed. After approximately 30 seconds, bleeding at each gingival unit will be recorded according to the following scale: 0 (Absence of bleeding after 30 seconds); 1 (Bleeding after 30 seconds); 2 (Immediate bleeding).

CONTACTS AND LOCATIONS:
Overall Officials: Chhaju Ram Goyal, DDS, Principal Investigator — All Sum Research Center Ltd.
Locations (1):
- All Sum Research Center Ltd.; 6635 Kitimat Road, Units 36 & 37, Mississauga, Ontario, Canada, Canada

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Araujo MWB, Charles CA, Weinstein RB, McGuire JA, Parikh-Das AM, Du Q, Zhang J, Berlin JA, Gunsolley JC. Meta-analysis of the effect of an essential oil-containing mouthrinse on gingivitis and plaque. J Am Dent Assoc. 2015 Aug;146(8):610-622. doi: 10.1016/j.adaj.2015.02.011. PMID 26227646
- [Background] Lobene RR, Weatherford T, Ross NM, Lamm RA, Menaker L. A modified gingival index for use in clinical trials. Clin Prev Dent. 1986 Jan-Feb;8(1):3-6. No abstract available. PMID 3485495
- [Background] Saxton CA, van der Ouderaa FJ. The effect of a dentifrice containing zinc citrate and Triclosan on developing gingivitis. J Periodontal Res. 1989 Jan;24(1):75-80. doi: 10.1111/j.1600-0765.1989.tb00860.x. PMID 2524573
- [Background] Van der Weijden GA, Timmerman MF, Nijboer A, Reijerse E, Van der Velden U. Comparison of different approaches to assess bleeding on probing as indicators of gingivitis. J Clin Periodontol. 1994 Oct;21(9):589-94. doi: 10.1111/j.1600-051x.1994.tb00748.x. PMID 7806674
- [Background] CHILTON NW. Studies in the design and analysis of dental experiments. II. A four-way analysis of variance. J Dent Res. 1960 Mar-Apr;39:344-60. doi: 10.1177/00220345600390021601. No abstract available. PMID 13809868
- [Background] Newman, MG, Takei, H, Klokkevold, PR, Carranza, FA; 2018; Newman and Carranza's Clinical Periodontology E-Book, 13th Edition; Saunders; p.387
- [Background] Turesky S, Gilmore ND, Glickman I. Reduced plaque formation by the chloromethyl analogue of victamine C. J Periodontol. 1970 Jan;41(1):41-3. doi: 10.1902/jop.1970.41.41.41. No abstract available. PMID 5264376
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CCSORC002549&attachmentIdentifier=780ba35c-fa01-403b-89d2-0afad13daf23&fileName=Infinity_2___CCSORC002549___Summary_CSR___Redacted.pdf&versionIdentifier=